CLINICAL TRIAL: NCT02828566
Title: Intranasal Ketamine Versus Intravenous Ketamine for Procedural Sedation in Children: a Multi-centre Randomized Controlled Non-inferiority Trial
Brief Title: Intranasal Ketamine for Procedural Sedation
Acronym: INK
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 106550
Record Dates: First submitted 2016-06-30; First posted 2016-07-11 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-03

CONDITIONS: Bone Fractures; Dislocations
MeSH Terms: conditions — Fractures, Bone; Joint Dislocations | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IN ketamine and IV saline (Experimental): Ketamine, single dose, 10 mg/kg (0.1 mL/kg) of 100 mg/mL solution delivered intranasally using an atomizer and divided to both nares to a maximum of 800 mg (8 mL) AND 0.9% normal saline (NS) 0.02 to 0.03 mL/kg delivered intravenously to a maximum of 2.4 mL
  Interventions: Drug: IN ketamine; Drug: IV saline 0.9%
- IV ketamine and IN saline (Active Comparator): Ketamine, single dose, 1 to 1.5 mg/kg (0.02 to 0.03 mL/kg) of 50 mg/mL solution delivered intravenously, to a maximum of 120 mg (2.4 mL) AND 0.9% normal saline (NS) 0.1 mL/kg delivered intranasally using an atomizer and divided to both nares, to a maximum of 8 mL
  Interventions: Drug: IV ketamine; Drug: IN saline 0.9%

INTERVENTIONS:
Drug: IN ketamine — Intranasal ketamine 100 mg/mL solution (10 mg/kg, maximum 800 mg)
  Other Names: ketamine hydrochloride
  Arms: IN ketamine and IV saline
Drug: IV ketamine — Intravenous ketamine 50 mg/mL solution (1 to 1.5 mg/kg, maximum 120 mg)
  Other Names: ketamine hydrochloride
  Arms: IV ketamine and IN saline
Drug: IN saline 0.9% — Intranasal 0.9% normal saline
  Arms: IV ketamine and IN saline
Drug: IV saline 0.9% — Intravenous 0.9% normal saline
  Arms: IN ketamine and IV saline

SUMMARY:
This study will examine the effectiveness of intranasal (IN) ketamine compared to standard intravenous (IV) ketamine administration for simple reductions of orthopaedic injuries in the paediatric population. The aim is to assess if IN administration is equivalent to the current standard of care, IV. The population to be studied is children 4-17 years of age who require a simple orthopaedic reduction. Following a double dummy approach to overcome the difficulty in masking interventions, each participant will receive both IV and IN interventions, only one of which will be the real drug. Procedural sedation and analgesia (PSA) will be assessed using the Dartmouth Operative Conditions Scale (DOCS).

DETAILED DESCRIPTION:
Randomization and concealment of allocation will be pharmacy-controlled using a computerized central randomization service. The treating physician, bedside nurse, research assistant, and participant will be blinded to the intervention. Eligible participants will be randomized in a 1:1 allocation ratio with a stratified block design of four or six to either (1) IN ketamine (each single dose, 10 mg/kg prepared in 0.9% NS in 3 mL syringe and atomizer, to a maximum of 8 mL) PLUS IV 0.9% NS 0.02 mL/kg or (2) IV ketamine (single dose, 1 mg/kg, to a maximum 80 mg) PLUS intranasal 0.9% NS 0.10 mL/kg divided to both nares. Due to the perceptible differences in interventional routes, each participant will receive both IV and IN interventions using this double-dummy approach. For IN dose volumes less than or equal to 0.5 mL, the entire dose will be delivered into 1 nostril and for doses greater than 0.5 mL, the dose will be divided equally between both nares. Adjunctive sedation will be given as needed in the form of IV ketamine, any dose, for participants who are adequately sedated 1 minute after IV administration at the discretion of the treating physician. Inadequate sedation in this context refers to one of the following: participant's vocalizations are consistent with pain OR participant withdraws or localizes due to pain. Eligible participants will be identified by the treating physician after viewing the radiographs and performing a clinical assessment. The physician will then inform a research assistant (RA) that the participant is eligible. The RA will then seek informed consent and explain the protocol to the family. Baseline demographic information will be obtained. Informed consent for PSA and a pre-anesthetic assessment will be performed by the treating physician in accordance with the usual standard of care. The RA will record a continuous video of the participant's entire body and monitor using an iPad starting immediately after the IV intervention until the participant is awake and able to tolerate oral fluids. DOCS scores will be obtained by two trained outcome assessors every 30 seconds for the entire duration of the video. The outcome assessors will also score the entire video for emergence delirium using the Paediatric Anesthesia Emergence Delirium (PAED) scale every 5 minutes beginning at the completion of fracture reduction until the participant is awake and drinking. Participants will receive standard monitoring of oxygen saturation, blood pressure, respiratory rate, apnea, heart rate, and rash by the attending nurse and physician every 5 minutes as per the usual standard of care. The usual standard of care also includes monitoring post-anesthetic for the presence of known idiosyncratic effects of ketamine that include vomiting, seizure, headache, emergence reaction, and hypersensitivity. The RA will obtain this information from the nursing record at discharge and based on consensus-based Canadian recommendations. Immediately prior to discharge, the RA will also record the duration of stay in the ED, parental, patient, and physician satisfaction with PSA using a 5-item Likert scale, and nasal irritation

ELIGIBILITY:
Inclusion Criteria:

1. Age 4 -17 years
2. Up to 80 kg
3. Presenting the paediatric emergency department
4. Require a closed reduction by procedural sedation and analgesia
5. Acute (=< 48 hours) distal radius and/or ulna fracture that is angulated with or without displacement
6. No more than 0.5 cm shortening in either the radius or ulna (not both)

Exclusion Criteria:

1. Previous hypersensitivity reaction to ketamine
2. Globe rupture
3. Traumatic brain injury with intracranial hemorrhage
4. History of uncontrolled hypertension
5. Nasal bone deformity
6. Duration of reduction expected to be greater than 20 minutes
7. Poor English or French fluency in the absence of a native language interpreter
8. American Society of Anesthesiologists (ASA) class of 3 or greater
9. Previous sedation with ketamine within 24 hours
10. Previous diagnosis of schizophrenia or psychosis based on DSM-V criteria
11. Pregnancy
12. Neuro-cognitive impairment that precludes informed consent, assent, or ability to self-report pain and satisfaction
13. Multi-limb trauma
14. Hemodynamic compromise
15. Glasgow coma score < 15
16. Fracture is comminuted
17. Fracture is associated with a dislocation
18. Hematoma block at index visit
19. Unilateral or bilateral nasal obstruction (due to infectious or allergic rhinitis, nasal polyps, septal hematoma, or septal deviation)

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 470 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Adequacy of sedation | Duration of fracture reduction
  Proportion with DOCS score -2 to +2 for duration of fracture reduction

SECONDARY OUTCOMES:
Depth of sedation | Duration of fracture reduction
  Score using Pediatric Sedation State Scale
Onset of adequate sedation | Within 1 hour following intervention
  Time interval from first IN sprays to first DOCS score between -2 and +2 in minutes
Duration of sedation | Within 2 hours following intervention
  Duration of time between the first DOCS score -2 to +2 to last DOCS score between -2 and +2 post-fracture reduction
Proportion of time participant adequately sedated during fracture reduction | Within 2 hours following intervention
  Proportion of time DOCS score is -2 to +2 during fracture reduction.
Adverse events | Within 2 hours following intervention
  The proportion of participants with adverse effects between groups will be compared. The list of adverse effects was chosen based on known adverse effects associated with ketamine and consensus-based recommendations for reporting for procedural sedation and analgesia in children.
Length of stay due to PSA | Within 3 hours of intervention
  Time interval from the first pair of IN sprays to discharge
Duration of procedure | Within 3 hours of intervention
  Time of the first pair of IN sprays to the end of cast or splint application
Caregiver satisfaction | Within 2 hours of intervention
  Obtained when patient is awake and drinking using a Visual Analog Scale; Parents not wishing to remain in proximity of child for sedation may opt out
Participant satisfaction | Within 2 hours of intervention
  Obtained when patient is awake and drinking using a Visual Analog Scale; Satisfaction will only be assessed in children at least eight years of age as the VAS has not been validated in younger children.
Physician satisfaction | Within 2 hours of intervention
  Obtained immediately prior to discharge using a Visual Analog Scale
Nurse satisfaction | Within 2 hours of intervention
  Obtained immediately prior to discharge using a Visual Analog Scale
Requirement for additional sedative medication | Within 2 hours of intervention
  Number of doses and type of adjunctive sedative medication required; Deemed inadequate if additional sedative medication given (for IN ketamine group only)
Analgesic medication | Within 2 hours of intervention
  Number of doses and type of analgesic medication required
Pain | Within 2 hours of intervention
  Pain scores will be recorded using the FPS-R on arrival and when the child is awake and drinking
Emergence delirium | 20 to 80 minutes post-IV intervention
  The proportion of children experiencing emergence delirium will be compared using the Paediatric Anesthesia Emergence Delirium (PAED) scale scored from the video every 5 minutes by an outcome assessor starting when fracture reduction is complete to when awake and drinking
Nasal irritation | Within 2 hours following intervention
  Measured using the Faces Pain Scale - Revised when awake and drinking
Successful sedation | Within 2 hours following intervention
  Successful sedation - Based on the definition of Bhatt et al., this will be defined as no unpleasant patient recall of the procedure, no resistance or restraint required during the procedure, no permanent sedation-related complication or no sedation-related event requiring abandonment of the procedure.
  Defined as: no unpleasant patient recall of the procedure, no resistance or restraint required during the procedure, no permanent sedation-related complication or no sedation-related event requiring abandonment of the procedure.
  Defined as no unpleasant recall of procedure, no resistance or restraint, no permanent sedation related complication, no sedation-related event requiring abandonment of procedure
Adjunctive IV therapy | Within 2 hours following intervention
  Other reasons for IV insertion (analgesia, anxiolysis, fluids, etc.)
Number of IN sprays received / Intended number of sprays | Within 2 hours following intervention
  Number of IN sprays received / Intended number of sprays
Number of IV attempts | Within 2 hours following intervention
  Number of IV attempts and time to IV insertion Number of IV attempts
Time to IV insertion | Within 2 hours following intervention
  Time from first breakage of skin to establishment of successful flow with a flush

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Poonai, MD, Principal Investigator — Western University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heath A, Offringa M, Pechlivanoglou P, Rios JD, Klassen TP, Poonai N, Pullenayegum E; KidsCAN PERC Innovative Paediatric Clinical Trials Team. Determining a Bayesian predictive power stopping rule for futility in a non-inferiority trial with binary outcomes. Contemp Clin Trials Commun. 2020 Apr 8;18:100561. doi: 10.1016/j.conctc.2020.100561. eCollection 2020 Jun. PMID 32300671